CLINICAL TRIAL: NCT04304170
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial of the Effect of Dietary Supplementation With Bifidobacteria and Fructo-oligosaccharides (FOS) on Bowel Movement Frequency and Intestinal Biological Markers in Seniors Presenting Slowed Intestinal Transit
Brief Title: Dietary Supplementation Effects on Bowel Movement Frequency and Intestinal Biological Markers in Seniors Presenting Slowed Intestinal Transit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: Vesale Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1487
Record Dates: First submitted 2020-02-26; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Constipation
Keywords: Constipation; Probiotic; Prebiotic
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: For each subject enrolled in the trial, the planned length of the trial was 44 days composed of a 14 day period at the beginning of the study without taking the trial product and a 30 day period when it was taken. The trial included three visits to the CEN Experimental Centre at D-14, D0 and D30. The product was taken from D1 onwards, the day after the enrolment visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum group (Experimental): The dietary supplement under study was composed of fructo-oligosaccharides - FOS: 4.95 gr / sachet and Bifidobacterium animalis lactis: VES002 (LMG P-28149): 5 billion / sachet. They came in the form of sachets of powder to be diluted in a glass of water. Doses were 2 sachets per day for the first 5 days and then 1 sachet per day for the next 25 days.
  Interventions: Dietary Supplement: VES002
- Placebo group (Placebo Comparator): The comparative product was a placebo that looked strictly identical to the verum and contained only excipients (60% maltodextrin / 40% sucrose).They came in the form of sachets of powder to be diluted in a glass of water. Doses were 2 sachets per day for the first 5 days and then 1 sachet per day for the next 25 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: VES002 — The sachets were to be dissolved in 200 ml of water at room temperature to be taken before breakfast.
  Arms: Verum group
Other: Placebo — The sachets were to be dissolved in 200 ml of water at room temperature to be taken before breakfast.
  Arms: Placebo group

SUMMARY:
This randomized, double-blind, controlled clinical trial among healthy volunteers with infrequent bowel movements but not severe constipation evaluate the effects of a supplementation in "symbiotic" on intestinal transit of subjects with few bowel movements per week with a verum group treated with a dietary supplement composed of fructo-oligosaccharides - FOS: 4.95 gr / sachet and Bifidobacterium animalis lactis: VES002 (LMG P-28149): 5 billion / sachet and a placebo group treated with a comparative product hat looked strictly identical to the verum and contained only excipients (60% maltodextrin / 40% sucrose).

The claim investigated corresponds to the section of the new EFSA (European Food Safety Authority) guidance of 2016 entitled "Claims on maintenance of normal defecation".

DETAILED DESCRIPTION:
Few studies have been made in France of the epidemiology of constipation although it is a frequent reason for visits to the doctor or for seeking advice from pharmacists. The prevalence of constipation in European and North American populations is reportedly of the order of 15% on average and it is 2.2 times more frequent among women than men. Hammond and Harari show there is an increased frequency of constipation from the age of 50 years onwards and that it substantially impacts quality of life. This can be explained in part by significant changes in the workings of the gastro-intestinal system in the course of normal ageing with reduced numbers of bifidobacteria in the gut.

These disorders are a major reason for taking oral and local drugs that are not without their side-effects and entail substantial healthcare costs. lifestyle rules combining appropriate fluid intake, regular physical activity and a high-fibre diet should be systematically recommended to such patients. "Symbiotic" dietary supplements combining probiotics and prebiotics may also be recommended provided that their effects have been properly validated. The symbiotic combination proposed in this clinical study is made up of fructo-oligosaccharides (FOS) sold as Actilight FOS (Beghin Say) and bifidobacteria BB12. Each of these components has been the subject of numerous studies showing improved intestinal transit especially in the elderly. A recent meta-analysis of the main studies published in Medline, Embase and The Cochrane Library has concluded that symbiotic with FOS and probiotics have a positive effect on bowel movement frequency and stool consistency.

The change in European regulations requires that clinical studies be conducted to secure EFSA claims for these dietary supplements. Such studies should also show an objective clinical benefit and factors such as a dose-dependent effect and/or the modification of biological markers that might confirm any such positive effect.

This randomized, double-blind, controlled clinical trial among healthy volunteers with infrequent bowel movements but not severe constipation serves this purpose. The claim investigated corresponds to the section of the new EFSA guidance of 2016 entitled "Claims on maintenance of normal defecation".

The primary endpoint of this trial is to evaluate the effect of supplementation in symbiotic on intestinal transit of subjects with few bowel movements per week.

The secondary endpoints are to evaluate:

* both clinical criteria such as changes in stool appearance, quality of life and mood, relief and satisfaction of participants;
* and biological criteria such as changes in markers of gut function, low-grade chronic inflammation markers and gut microbiota markers.

The safety of product use and compliance are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female volunteers aged 50-70 years with ≥1 and ≤3 bowel movements per week in the month before the selection visit and in the two weeks before the enrolment visit,
* at least one in four bowel movements had to involve hard faeces or separate lumps of faeces (Bristol scale class 1) in the three months before enrolment.

Exclusion Criteria:

* subjects who, in the 30 days before the selection visit or at the time of the visit, had taken drugs, dietary supplements or any foodstuff enhanced in or containing substances, bacteria or yeasts and that might have an effect on the gut and more specifically on intestinal transit, digestive comfort, production of gas, or the occurrence of abdominal pain. Such products were also prohibited throughout the study. The same applied to subjects on a particular diet (vegetarian, vegan, hyper-protein, etc.), a low-calorie diet or under medical treatment which in the investigator's view might interfere with the evaluation of the study criteria (antibiotics, corticoids, anticholinergics, antidepressants, antiemetics, diuretics, calcium channel blockers, antiparkinson drugs, antipsychotics, antacids, analgesics, NSAIDS, H2 receptor antagonists, hypnotics, sedatives, iron supplements, opioids and narcotics, laxatives, anti-diarrhoeal drugs, anti-reflux drugs, etc.),
* subjects who drink more than three glasses of wine a day or two 25 cl glasses of beer a day, or one glass of spirits per day and those who drink more than five cups of coffee per day;
* subjects with a body mass index (BMI) of more than 30,
* subjects with type I or II diabetes,
* subjects with constipation attributable to an organic or anatomical cause;
* subjects with a history of chronic or inflammatory gastro-intestinal disease;
* subjects with a history of digestive tract operation and especially bariatric surgery;
* subjects with a fibre intake exceeding the recommended levels (more than six portions of fruit and vegetables per day according to the PNNS - national nutrition and health programme - questionnaire) or engaging in intense sport for more than 10 hours per week.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in intestinal transit | Reported daily from Day -14 to Day 30
  Evaluated by the frequency of bowel movements

SECONDARY OUTCOMES:
Changes in stool aspect | Reported daily from Day -14 to Day 30
  Evaluated by the Bristol Stool Form Scale (BSFS) ; The BSFS classifies stools into seven categories, including type 1, separate hard lumps, like nuts; type 2, sausage-shaped, but lumpy; type 3, like a sausage but with cracks on the surface; type 4, like a sausage or snake, smooth and soft; type 5, soft blobs with clear-cut edges; type 6, fluffy pieces with ragged edges, a mushy stool; type 7, watery, no solid pieces [25]. These types are categorized into slow transit (types 1 and 2), normal transit (types 3-5), and fast transit (types 6 and 7).
Changes in quality of life | Day -14 to Day 30
  Evaluated by the quality of life questionnaire SF(Short Form) 12 consisting of 12 questions relating to: physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations and general mental health (psychological distress and psychological well-being). This instrument yields two summary scores: a Mental Component Score from 19 (poor mental condition) to 56 (excellent mental condition) and a Physical Component Score (PCS) from 24 (poor physical condition) to 56 (excellent physical condition).
Mood changes | Reported daily from Day-14 to Day 30
  Evaluated by the Brief Mood Introspection Scale (BMIS) consisting of 16 mood adjectives (Lively, Drowsy, Happy, Grouchy, Sad, Peppy, Tired, Nervous, Caring, Calm, Content, Loving, Gloomy, fed up, Jittery, Active). Subjects were asked to circle the phrases describing their present mood (with XX = definitely do not feel; X = do not feel; V = slightly feel; VV = definitely feel on the diverse adjectives). The BMIS was scored for Pleasant-Unpleasant Mood, Arousal-Calm Mood, Positive-Tired Mood and Negative-Relaxed Mood according to the Mayer's method.
Relief of subjects | At Day 30
  Evaluated on the PGI-I (Patient Global Impression of Improvement) scale; The PGI-I is a 1-item questionnaire asking to rate the perceived change in his/her condition in response to therapy from 1 (Very much better) to 7 (Very much worse)
Satisfaction toward treatment | At Day 30
  Evaluated on a 5 points Likert scale (0 : very unsatisfied ; 5 : very satisfied)
Tolerance: occurrence of diarrhoea | At Day 30
  Evaluated especially by the occurrence of diarrhoea

OTHER OUTCOMES:
Plasma peptides | At Day -7 and Day 30
  Plasma concentrations of pancreatic polypeptide (PP), glucose-dependent insulinotropic peptide (GIP), leptin, ghrelin, insulin
Gut microbiota analyses | At Day -7 and Day 30
  PCR (Polymerase Chain Reaction) and metagenomic analysis of bacteria taxa on faecal samples
Low-grade inflammation plasma markers | At Day -7 and Day 30
  Plasma concentrations of cytokines, interleukins, monocyte chemotactic protein-1, interferon and tumor necrosis factor
Safety plasma parameters | At Day -14 and Day 30
  Plasma concentrations of lipids (Chlolesterol, triglycerides), blood count, glycaemia, alanine aminotransferase, aspartate aminotransferase

CONTACTS AND LOCATIONS:
Locations (1):
- CEN Nutriment, Dijon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No